CLINICAL TRIAL: NCT00475436
Title: A Single-centre, Randomised, Double-blind, Placebo-controlled, Dose-ascending, 3-cohort Parallel-group Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of GSK573719 Administered as Singledoses (750 μg and 1000 μg) and Repeat Doses Over 14 Days (250 μg-1000 μg Once-daily) of GSK573719 in Healthy Male and Female Subjects.
Brief Title: A Single Centre Randomized Study Evaluating The Safety And Tolerability Of GSK573719 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AC4106889
Record Dates: First submitted 2007-05-16; First posted 2007-05-21 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: muscarinic receptor antagonist; GSK573719,; chronic obstructive pulmonary disease,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — GSK573719

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: GSK573719

INTERVENTIONS:
Drug: GSK573719

SUMMARY:
GSK573719 is a high-affinity specific muscarinic receptor (mAChR) antagonist which is being developed for once daily treatment of chronic obstructive pulmonary disease (COPD). The long duration of action of GSK573719 when administered via inhalation in animal models supports the potential for use as a once-daily bronchodilator for COPD

DETAILED DESCRIPTION:
A single-centre, randomised, double-blind, placebo-controlled, dose-ascending, 3-cohort parallel-group study to evaluate the safety, tolerability, pharmacodynamics and pharmacokinetics of GSK573719 administered as single doses (750µg and 1000µg) and repeat doses over 14 days (250µg-1000µg once-daily) of GSK573719 in healthy male and female subjects

ELIGIBILITY:
Inclusion criteria:

* Healthy Caucasian male subjects or healthy Caucasian female subjects of non-childbearing potential
* Aged between 18-55 years
* Non-smokers
* Normal spirometry (FEV1 = 80% of predicted, FEV1/FVC = 70%)
* A signed and dated written informed consent is obtained from the subject
* The subject is capable of giving informed consent
* Available to complete the study
* Subject has a BMI within the range 18.0-30.0kg/m2 inclusive

Exclusion criteria:

* Any clinically important abnormality identified at the screening medical assessment
* A history of breathing problems
* A mean QTc(B) value at screening >450msec, the QTc(B) of all 3 screening ECGs are not within 10% of the mean, or an ECG that is not suitable for QT measurements
* A history of elevated resting blood pressure or a mean blood pressure equal to or higher than 140/90 mmHg at screening
* A mean heart rate outside the range 40-90 bpm at screening
* History of use of tobacco products within 6 months of screening, or positive urine cotinine at screening
* Subjects with a 2D6 poor metabolizer genotype (Caucasian)
* The subject has donated a unit (400ml) of blood within 60 days of screening, or, intends to donate during the study
* The subject is currently taking regular (or course of) medication, whether prescribed or not
* The subject has taken prescription medications within the past 2 weeks prior to dosing or OTC medications within 48 hours prior to dosing
* The subject has participated in a study with a new molecular entity or any other trial within a period of 3 months prior to dosing
* The subject has tested positive for hepatitis C antibody, hepatitis B surface antigen or HIV
* The subject has a positive pre-study drug screen
* The subject has a positive pre-study alcohol screen
* The subject has a suspected history of alcohol abuse within the six months previous to the screening visit
* The subject is unable to use the DISKUS
* The subject has a known allergy or hypersensitivity to ipratropium bromide, atropine and any of its derivatives
* The subject has a known allergy or hypersensitivity to milk protein or the excipient lactose monohydrate
* Subjects who might have prostatic hypertrophy, bladder outlet obstruction, or narrow angle glaucoma

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2007-05-14 (Actual); Primary Completion 2007-09-18 (Actual); Study Completion 2007-09-18 (Actual)

PRIMARY OUTCOMES:
General safety and tolerability endpoints: adverse events, blood pressure, heart rate, 12-lead ECG, Holter and Lead II ECG monitoring, lung function and clinical laboratory safety tests throughout the study | throughout the study

SECONDARY OUTCOMES:
- Ambulatory blood pressure for repeat dosing - 24hr Holter monitoring for repeat dosing - Plasma and urine concentrations of GSK573719 and derived pharmacokinetic parameters | throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Cahn A, Tal-Singer R, Pouliquen IJ, Mehta R, Preece A, Hardes K, Crater G, Deans A. Safety, tolerability, pharmacokinetics and pharmacodynamics of single and repeat inhaled doses of umeclidinium in healthy subjects: two randomized studies. Clin Drug Investig. 2013 Jul;33(7):477-88. doi: 10.1007/s40261-013-0088-7. PMID 23784369
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study AC4106889 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/AC4106889?search=study&search_terms=AC4106889#rs
- Available data/document: Dataset Specification: AC4106889 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: AC4106889 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: AC4106889 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: AC4106889 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: AC4106889 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: AC4106889 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: AC4106889 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register